CLINICAL TRIAL: NCT01832610
Title: A Multi Center, Post Approval Study Providing Continued Evaluation and Follow-up on Patients Who Received a HeartWare® Ventricular Assist System During IDE Trials for the Treatment of Advanced Heart Failure
Brief Title: Post- Approval Study on Patients Who Received a HeartWare HVAD® During IDE Trials
Acronym: HW-PAS-03
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: HW-PAS-03
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HeartWare® VAS: Ventricular Assist Device (HeartWare® VAS)
  Interventions: Device: HeartWare® VAS

INTERVENTIONS:
Device: HeartWare® VAS — The HeartWare® LVAD is an implantable centrifugal pump that was designed to provide flows up to 10 L/min in a small device which is both lightweight and simple to use.
  Other Names: HVAD®

SUMMARY:
Patients will be approached to participate in this PAS after the HeartWare® Ventricular Assist System receives PMA approval for the indicated use as a bridge to cardiac transplantation.

DETAILED DESCRIPTION:
Patients who participated in prior trials will be approached for this PAS as follows:

* Patients who are on continued HeartWare® System support, (original or exchange device)
* Patients who have been explanted for transplant or recovery and have not yet completed 6 months of follow-up

Patients who participated in prior trials who will not be approached to participate in this follow-up study include:

• Patients who have been explanted for transplant or recovery and have completed at least 6 months of follow-up (documented in the prior IDE trial).

No new patients are being screened or implanted with the HeartWare® System for this trial, it is a follow-up trial only.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has participated in a prior HeartWare trial under IDE G070199.
2. The patient was implanted with the HeartWare® Ventricular Assist System and was an active patient in the prior trial.
3. The patient has signed informed consent for participation in the study.

Exclusion Criteria:

1. The patient is unwilling or unable to comply with trial requirements.
2. The patient did not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population consists of patients who were at risk of death from refractory, advanced heart failure and implanted with a HeartWare® Ventricular Assist System under IDE G070199.
  Patients must have participated as a study patient in a prior HeartWare trial under IDE G070199, and been implanted with the HeartWare® System
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Stanford University School of Medicine, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida - Gainesville, Gainesville, Florida
  - University of Miami / Jackson Memorial Hospital, Miami, Florida
  - The Emory Clinic Inc., Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - IU Health Methodist, Indianapolis, Indiana
  - Jewish Hospital - Rudd Heart and Lung Institute, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University / Barnes Jewish Hospital, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas - South Western, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - Northwest Cardiothoracic &Transplant Surgeons, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 101 enrolled subjects, 17 subjects enrolled post-transplant and were no longer on the HVAD device at the time of enrollment, leaving 84 subjects who enrolled while still on the HVAD device.
Period: Overall Study
Arm/Group | HeartWare® VAS
Started | 101
Completed | 97
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: All enrolled subjects are included.
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment into HW-PAS-03
  years | 54.4 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Black or African American | 37
  Native Hawaiian or Other Pacific Islander | 1
  White | 59
  Other | 3
Enrollment Characteristics [Count of Participants; unit: Participants]
  On Device | 84
  Post Transplant | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival on Device
Description: Overall survival is the probability (expressed as a percent of 100) the participant did not die within 5 years post implant via the Kaplan-Meier method. Participants that did not die were censored at the time of last follow-up or their end of study at 5 years post implant, whichever occurred first.
Time Frame: Implant to 5 years
Population: All enrolled subjects are included
Measure: Number; unit: Percent Probability of Survival
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 101
Percent Probability of Survival | 52.9

2. Secondary Outcome: Final Patient Status
Description: The number and percentage of participants with a given outcome (e.g., alive on device, transplant, death, etc.) as of their last follow up or end of study, whichever occurred first.
Time Frame: Implant to 5 years
Population: All enrolled subjects are included.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 101
Participants
  Alive on Original Device | 21
  Alive Post Exchange | 5
  Alive Post Explant for Transplant | 41
  Alive Post Explant for Recovery | 0
  Dead on Original Device | 22
  Dead Post Exchange | 6
  Dead Post Explant for Transplant | 6
  Dead Post Explant for Recovery | 0

3. Secondary Outcome: Re-hospitalizations
Description: A summary of the number of re-hospitalizations per participant from enrollment into HW-PAS-03 throughout their participation in the study.
Time Frame: Enrollment into HW-PAS-03 to 5 years
Population: Participants who enrolled into the trial on device are included.
Measure: Mean (Standard Deviation); unit: Re-hospitalizations
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 84
Re-hospitalizations | 3.9 (3.80)

4. Secondary Outcome: Number of Participants Experiencing Any Adverse Event Per Intermacs Definition
Description: Number of participants with an Intermacs adverse event, per the Intermacs definitions. An adverse event is any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in participants, users or other persons whether or not related to the medical device.
Time Frame: Enrollment into HW-PAS-03 to 5 years
Population: Participants who enrolled into the trial on device are included.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 84
Participants | 66

5. Secondary Outcome: Health Status Change Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Health Status change as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score. The KCCQ is a disease-specific patient-reported outcomes measure for patients with heart failure. It consists of 23 items, is comprised of 7 clinically relevant scales (Symptom Frequency, Symptom Burden, Symptom Stability, Physical Limitation, Social Limitation, Quality of Life, and Self-Efficacy), and yields 3 summary scores (Clinical Summary, Total Symptom, and Overall Summary Scores). Scale and summary scores range between 0 and 100, with higher scores indicating better health status (e.g., better functioning, fewer symptoms, better quality of life). The Overall Summary Score is calculated as the mean of the Physical Limitation, Total Symptom, Quality of Life and Social Limitation scores. A positive change in score from baseline indicates an improvement.
Time Frame: Change from baseline to 5 years
Population: Participants who enrolled into the trial on device are included. Participants also had to reach the Month 60 visit and complete both the baseline and Month 60 assessments to be analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 15
score on a scale | 20.1 (21.32)

6. Secondary Outcome: Health Status Change Measured by EuroQol EQ-5D (Version 5L)
Description: The EuroQol-5D (version 5L) is a brief self-administered, validated instrument consisting of 2 parts. The second part consists of the EQ-5D general health status as measured by a visual analog scale (EQ-5D VAS). EQ-5D VAS measures the participant's self-rated health status on a scale from 0 (worse imaginable health state) to 100 (best imaginable health state).
Time Frame: Enrollment to 5 years
Population: Participants who enrolled into the trial on device are included. Participants also had to reach the Month 60 visit complete the assessment to be analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 19
score on a scale | 66.84 (22.124)

7. Secondary Outcome: Change in Functional Status Measured by New York Heart Association (NYHA) Class
Description: Change in Functional status, as measured by New York Heart Association (NYHA) class. There are 4 levels of NYHA:
  I (Mild): No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea.
  II (Mild): Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
  III (Moderate): Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV (Severe): Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
  Improvement is defined as moving from a higher numerical NYHA level to a lower numerical NYHA level (e.g., IV to III).
Time Frame: Change from baseline to 5 years
Population: Participants who enrolled into the trial on device were included. Participants also had to reach the Month 60 visit and complete the assessment to be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 22
Participants
  No Change in NYHA Class | 2
  Improved 1 NYHA Class | 5
  Improved 2 NYHA Classes | 7
  Improved 3 NYHA Classes | 8

8. Secondary Outcome: Change in Functional Status Measured by 6-minute Walk
Description: Change in functional status, as measured by 6-minute walk test. A positive change in score from baseline indicates an improvement.
Time Frame: Change from baseline to 5 years
Population: Participants who enrolled into the trial on device are included. Subjects also had to reach the Month 60 visit and complete the assessment or indicate Not Completed to be analyzed at both the baseline and Month 60 visits. If the subject did not complete the assessment, a value of 0 was imputed.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 22
Meters | 106.6 (184.05)

ADVERSE EVENTS:
Time Frame: The adverse events are summarized from the date of enrollment through 5 years while on the originally implanted device. Only participants who enrolled into the trial on device are included.
Description: The Interagency Registry for Mechanically Assisted Circulatory Support (Intermacs) adverse event definitions are geared towards subjects who have a mechanical circulatory support device. Subjects who enrolled into the trial post-transplant (off device) (N=17) did not have any adverse events collected during the trial.
Arm/Group | HeartWare® VAS
All-Cause Mortality (participants affected / at risk) | 34/101
Serious Adverse Events (participants affected / at risk) | 62/84
Other Adverse Events (participants affected / at risk) | 10/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartWare® VAS (N=84)
Major Bleeding (Blood and lymphatic system disorders) | 19 (35)
Cardiac Arrhythmia (Cardiac disorders) | 12 (15)
Device Malfunction (Product Issues) | 29 (34)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hepatic Dysfunction (Hepatobiliary disorders) | 2 (3)
Hypertension (Cardiac disorders) | 1 (3)
Major Infection (Infections and infestations) | 37 (69)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Neurological Dysfunction (Nervous system disorders) | 14 (19)
Pericardial Fluid Collection (Cardiac disorders) | 0 (0)
Psychiatric Episode (Psychiatric disorders) | 5 (5)
Renal Dysfunction (Renal and urinary disorders) | 7 (7)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Right Heart Failure (Cardiac disorders) | 3 (3)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 1 (1)
Venous Thromboembolism (Vascular disorders) | 3 (3)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0)
Other Intermacs (General disorders) | 48 (161)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartWare® VAS (N=84)
Device Malfunction (Product Issues) | 5 (5)
Major Infection (Infections and infestations) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, the contract allows the principal investigator to publish their data after the release of the multi-center publication (or one year after the conclusion of the study if no multi-center publication is submitted) following the sponsor review for (a) disclosure of confidential information, and (b) information that would impair the sponsor's ability to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2013-09-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT01832610/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT01832610/SAP_001.pdf